CLINICAL TRIAL: NCT00564850
Title: Phase III, Multicentre, Non-comparative, Open and Single Stage Study to Assess the Efficacy and Safety of Pamoate of Triptorelin 11.25 MG in Children With Precocious Puberty
Brief Title: Efficacy and Safety Study of Pamoate of Triptorelin in Children With Precocious Puberty
Acronym: DECAPUB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2-54-52014-143; 2005-005644-11 (EudraCT Number)
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Results first posted 2011-12-01 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Precocious Puberty
MeSH Terms: conditions — Puberty, Precocious | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triptorelin pamoate 11.25mg (Decapeptyl® SR) (Experimental)
  Interventions: Drug: Triptorelin pamoate 11.25mg (Decapeptyl® SR)

INTERVENTIONS:
Drug: Triptorelin pamoate 11.25mg (Decapeptyl® SR) — One intra muscular injection at day 1 and month 3.

SUMMARY:
The purpose of the study is to assess the efficacy of triptorelin 11.25 mg pamoate in the delay of premature onset of puberty in girls less than 9 years and boys less than 10 years. This is measured by assessing the proportion of children who have a suppressed Luteinizing Hormone (LH) response to Gonadotropin Releasing Hormone (GnRH) test performed 3 months after injection with triptorelin 11.25 mg.

ELIGIBILITY:
Inclusion Criteria in the screening phase:

* Onset of sex characteristics (Tanner method) breast development in girls or testicular enlargement in boys before the age of 8 years in girls and 9 years in boys.
* Weight ≥ 20 kg.

Inclusion Criteria in the treatment phase:

* Proven central precocious puberty defined as onset of sex characteristics development (according to Tanner method) diagnosed before the age of 8 years in girls and 9 years in boys.
* Age at evaluation less than 9 years for girls and 10 years for boys.
* A pubertal response of LH to GnRH test in both sexes (stimulated LH ≥ 5 IU/l).
* Difference Bone age (BA) (according to Greulich et Pyle method) - Chronological age (CA) > 1 year.
* Testosterone level ≥ 0.5 ng/ml in boys.

Exclusion Criteria:

* Patient with a peripheral precocious puberty: extrapituitary secretion of gonadotropins or gonadotropin-independent gonadal or adrenal sex steroids secretion.
* Patient with a cerebral tumour requiring a neurosurgery or cerebral irradiation.
* Patient with a Body Weight ≥ 125% of the ideal weight for the height and age (growth curves).
* The patient has received a previous treatment with a GnRH analogue, or medroxyprogesterone or cyproterone acetate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (18):
- France (18):
  - Hôpital Hotel-Dieu (CHU), Angers
  - Hôpital Saint-Jacques, Besançon
  - Medical Centre, Bordeaux
  - Hôpital du Bocage, Dijon
  - Hôpital Flaubert, Le Havre
  - Hôpital Jeanne de Flandre, Lille
  - Hôpital Debrousse, Lyon
  - Hôpital de la Timone Enfants, Marseille
  - Hôpital Archet 2, Nice
  - Hôpital Trousseau, Paris
  - Hôpital St-Vincent de Paul, Paris
  - Hôpital Necker - Enfants Malades, Paris
  - Hôpital Robert Debré, Paris
  - American Memorial Hospital, Reims
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Hautepierre, Strasbourg
  - Hôpital de la Gespe, Tarbes
  - Hôpital des Enfants, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 62 participants were screened, of which 37 met the study's entry criteria and received at least one dose of investigational medicinal product. 25 participants failed screening. Participants were recruited from October 2007 at 18 Hospital clinics across France.
Groups:
- Triptorelin Pamoate 11.25 mg: 11.25 mg triptorelin pamoate via intramuscular injection at baseline and month 3.
Period: Overall Study
Arm/Group | Triptorelin Pamoate 11.25 mg
Started | 37
Completed | 35
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.2 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 1
Region of Enrollment [Number; unit: participants]
  France | 37
Weight [Mean (Standard Deviation); unit: Kg] | 32.76 (7.36)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a GnRH-stimulated LH Level ≤3 IU/L
Time Frame: 3 months after the first injection of triptorelin pamoate 11.25 mg
Population: Analyses performed on:
  * Intention to Treat (ITT): all patients having received ≥1 injection. Any subject with missing data is considered a non-responder.
  * Modified ITT (mITT): all ITT patients with ≥ Month 3 post-baseline assessment of primary efficacy criterion.
  * Per Protocol (PP): all mITT patients without major protocol deviations.
Measure: Number; unit: participants
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 37
participants
  Yes [ITT (n=37)] | 31 [68.0 to 93.8]
  No [ITT (n=37)] | 6
  Yes [mITT (n=34)] | 31 [76.3 to 98.1]
  No [mITT (n=34)] | 3
  Yes [PP (n=32)] | 30 [79.2 to 99.2]
  No [PP (n=32)] | 2

2. Secondary Outcome: Number of Participants Whose Intravenous (i.v.) GnRH-stimulated LH Response Was ≤3 IU/L
Time Frame: Month 6
Population: Analysis was performed on Intention to Treat population (ITT) defined as all participants having received at least one injection of 11.25 mg triptorelin pamoate. "n" indicates the number of patients who had an assessment at the visit.
Measure: Number; unit: participants
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 37
participants
  Yes (n=37) | 32 [71.2 to 95.5]
  No (n=37) | 5

3. Secondary Outcome: Follicle Stimulating Hormone (FSH) Level Following GnRH Test
Time Frame: Screening, month 3 and 6
Population: Analysis was performed on the ITT population. 3 participants and 2 participants had missing data at month 3 and month 6 respectively.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 37
IU/L
  Screening (n=37) | 11.84 (3.23)
  Month 3 (n=34) | 2.26 (2.5)
  Month 6 (n=35) | 2.34 (1.65)

4. Secondary Outcome: Basal FSH Level
Time Frame: Month 0, 1, 2, 3, 4, 5, and 6
Population: Analysis was performed on the ITT population. 2 participants had missing data at month 1, 3, 4 and 6. 1 and 3 participants had missing data at month 2 and month 5 respectively.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 37
IU/L
  Month 0 (screening, n=37) | 4.13 (2.65)
  Month 1 (n=35) | 0.67 (0.53)
  Month 2 (n=36) | 1.07 (0.82)
  Month 3 (n=35) | 1.11 (0.73)
  Month 4 (n=35) | 0.78 (0.39)
  Month 5 (n=34) | 1.41 (2.09)
  Month 6 (n=35) | 1.36 (1.24)

5. Secondary Outcome: Basal LH Level
Time Frame: Month 0, 1, 2, 3, 4, 5 and 6
Population: Analysis was performed on ITT population. 2 participants had missing data at month 1, 3, 4 and 6. 1 and 3 participants had missing data at month 2 and month 5 respectively.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 37
IU/L
  Month 0 (screening, n=37) | 1.49 (1.78)
  Month 1 (n=35) | 0.42 (0.22)
  Month 2 (n=36) | 0.42 (0.31)
  Month 3 (n=35) | 0.43 (0.27)
  Month 4 (n=35) | 0.43 (0.23)
  Month 5 (n=34) | 0.48 (0.70)
  Month 6 (n=35) | 0.44 (0.42)

6. Secondary Outcome: Number of Girls With Oestradiol Levels ≤ 20 pg/ml
Time Frame: Month 0, 1, 2, 3, 4, 5 and 6
Population: Analysis was performed on female patients in the ITT population. 2 participants had missing data at month 1, 3, 4 and 6. 1 participant and 3 participants had missing data at month 2 and 5 respectively.
Measure: Number; unit: participants
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 36
participants
  Yes - month 0 (n=36) | 22
  No - month 0 (n=36) | 14
  Yes - month 1 (n=34) | 34 [89.7 to 99.9]
  No - month 1 (n=34) | 0
  Yes - month 2 (n=35) | 34 [85.1 to 99.9]
  No - month 2 (n=35) | 1
  Yes - month 3 (n=34) | 33 [84.7 to 99.9]
  No - month 3 (n=34) | 1
  Yes - month 4 (n=34) | 34 [89.7 to 100]
  No - month 4 (n=34) | 0
  Yes - month 5 (n=33) | 33 [89.4 to 100]
  No - month 5 (n=33) | 0
  Yes - month 6 (n=34) | 33 [84.7 to 99.9]
  No - month 6 (n=34) | 1

7. Secondary Outcome: Testosterone Level
Time Frame: Month 0, 3 and 6
Population: Testosterone level from the male patient in the ITT population.
Measure: Number; unit: ng/ml
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 1
ng/ml
  Month 0 (screening) | 2.0
  Month 3 | 0.12
  Month 6 | 0.16

8. Secondary Outcome: Number of Girls With Inhibin B Levels < 6 pg/ml
Time Frame: Month 0, 3 and 6
Population: Analysis was performed on female patients in the ITT population. 2 participants had missing data at month 3 and month 6.
Measure: Number; unit: participants
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 36
participants
  Yes - month 0 (screening, n=36) | 18
  No - month 0 (screening, n=36) | 18
  Yes - month 3 (n=34) | 33 [84.7 to 99.9]
  No - month 3 (n=34) | 1
  Yes - month 6 (n=34) | 32 [80.3 to 99.3]
  No - month 6 (n=34) | 2

9. Secondary Outcome: Change From Screening in Pubertal Stage (Tanner Method) at Month 6
Description: Pubertal stage (graded from 1 to 5 for penis and breast development, graded from 1 to 6 for pubic hair development) according to the Tanner method was collected. A low stage (i.e. 1) corresponds to a pre-pubertal stage and a high stage (i.e. 5 or 6) to an adult stage. Any increase of grade was defined as 'increased' and no change in grade or a reduced grade was defined as 'stabilised or reduced'.
Time Frame: Between screening and month 6
Population: Analysis was performed on the ITT population. 2 participants had missing data for pubic hair stage and breast stage.
Measure: Number; unit: participants
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 37
participants
  Pubic hair stage stabilised or reduced (n=35) | 30
  Pubic hair stage increased (n=35) | 5
  Breast stage stabilised or reduced (n=34) | 32
  Breast stage increased (n=34) | 2
  Penis stage stabilised or reduced (n=1) | 1
  Penis stage increased (n=1) | 0

10. Secondary Outcome: Height Standard Deviation Score (SDS)
Description: Standard deviation (SD) is a standard term used in growth studies and represents Standard Deviations calculated as the patient value minus the mean divided by the standard deviation. Standard Deviation Scores vary depending on the age and sex of the child.
Time Frame: Month 0, 3 and 6
Population: Analysis was performed on the ITT population. 2 participants had missing data at month 6.
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 37
SD score
  Month 0 (baseline, n=37) | 1.25 (1.14)
  Month 3 (n=37) | 1.32 (1.16)
  Month 6 (n=35) | 1.32 (1.16)

11. Secondary Outcome: Body Mass Index (BMI) SDS
Time Frame: Month 0, 3 and 6
Population: Analysis was performed on the ITT population. 1 and 2 participants had missing data at month 0 and month 6 respectively.
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 37
SD score
  Month 0 (baseline, n=36) | 0.58 (0.85)
  Month 3 (n=37) | 0.64 (0.89)
  Month 6 (n=35) | 0.60 (0.78)

12. Secondary Outcome: Change From Baseline in Growth Velocity (GV) SDS at Month 6
Description: Change from baseline of GV was calculated as: GV at month 6 - GV at baseline. GV SDS was calculated using SAS algorithm.
  Growth velocity during the study was calculated using the two height measures as: GV = (Height at baseline - Height at screening)*365/delay between two height measures.
Time Frame: Baseline and month 6
Population: Analysis was performed on the ITT population. If GV at screening was missing, the value was derived from data recorded between 5 to 19 months ago otherwise GV at screening was considered missing. 9 participants had missing data.
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 37
SD score | -1.95 (2.07)

13. Secondary Outcome: Difference Between Bone Age and Chronological Age
Description: Bone age was defined according to Greulich and Pyle method. Chronological age was calculated using the date of birth.
Time Frame: Month 0 and 6
Population: Analysis was performed on the ITT population. 33 participants were assessed. 4 participants had missing data at month 6.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 37
years
  Month 0 (screening, n=37) | 2.09 (0.91)
  Month 6 (n=33) | 2.02 (0.88)

14. Secondary Outcome: Uterine Length
Time Frame: Month 0, 3 and 6
Population: Analysis was performed on female patients in the ITT population. 2 participants had missing data at month 3 and 6.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 36
mm
  Month 0 (screening, n=35) | 37.6 (10.6)
  Month 3 (n=34) | 37.4 (8.2)
  Month 6 (n=34) | 36.8 (6.9)

15. Secondary Outcome: Triptorelin Plasma Levels
Time Frame: Month 1, 2, 3, 4, 5 and 6
Population: Analysis was performed on the Pharmacokinetics (PK) Valid population defined as all participants who received at least one injection of 11.25 mg triptorelin pamoate and had at least one PK assessment. 2 participants had data missing at month 1,3 and 6. 1, 3 and 4 participants had data missing at month 2, 4 and 5 respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 37
ng/mL
  Month 1 (n=35) | 0.187 (0.115)
  Month 2 (n=36) | 0.048 (0.023)
  Month 3 (n=35) | 0.034 (0.018)
  Month 4 (n=34) | 0.201 (0.120)
  Month 5 (n=33) | 0.045 (0.023)
  Month 6 (n=35) | 0.030 (0.017)

ADVERSE EVENTS:
Arm/Group | Triptorelin Pamoate 11.25 mg
Serious Adverse Events (participants affected / at risk) | 1/37
Other Adverse Events (participants affected / at risk) | 7/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin Pamoate 11.25 mg (N=37)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin Pamoate 11.25 mg (N=37)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Injection site pain (General disorders) | 2 (2)
Hot flush (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days